CLINICAL TRIAL: NCT00043498
Title: Health Effects of Early-Life Exposure to Urban Pollutants in Minority Children
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 8977-CP-001
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Asthma; Development
Keywords: Pollutants
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We collected maternal urine during the third trimester of pregnancy, maternal blood at delivery, umbilical cord blood, meconium, blood and urine from the child at ages 24, 36, and 60 months.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A molecular epidemiologic study of African American and Hispanic mothers and newborns to investigate the role of common urban pollutants on procarcinogenic and developmental damage.

DETAILED DESCRIPTION:
The major objective of the proposed research is to study the impact of early-life exposures to common urban pollutants on neurobehavioral development and asthma in a sample of children living in three low-income, minority communities of New York City (Central Harlem, Washington Heights and the South Bronx). Using a molecular epidemiologic approach with monitoring, biomarkers, and clinical assessments at serial time points, we will extend our study of African-American and Latina urban mothers and children in order to follow the cohort through child age 11 years to assess the longer-term impact of exposures on child health and developmental outcomes.

ELIGIBILITY:
Enrollment eligibility was restricted to nonsmoking pregnant women 18-35 years of age who self-identified as either African American or Dominican and who had resided in northern Manhattan or the South Bronx in New York City for at least 1 year before pregnancy. Women were excluded if they used illicit drugs, had diabetes, hypertension, or known HIV, or had their first prenatal visit after the 20th week of pregnancy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present study enrolled 727 African American and Latino (Dominican) mothers and their children. The African American and Latino (Dominican) women were initially enrolled into the parent CCCEH study during pregnancy. Caucasian women are not included because a central purpose of the research is to evaluate health outcomes in a high risk, minority population.
Sampling Method: Non-Probability Sample
Enrollment: 727 (Actual)
Dates: Start 1997-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral development | 1 to 12 years
Asthma | 2-12 years

CONTACTS AND LOCATIONS:
Overall Officials: Frederica P Perera, DrPH, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, 722 W 168th St, 12th Floor, New York, New York, United States

REFERENCES:
- [Derived] Widen EM, Whyatt RM, Hoepner LA, Ramirez-Carvey J, Oberfield SE, Hassoun A, Perera FP, Gallagher D, Rundle AG. Excessive gestational weight gain is associated with long-term body fat and weight retention at 7 y postpartum in African American and Dominican mothers with underweight, normal, and overweight prepregnancy BMI. Am J Clin Nutr. 2015 Dec;102(6):1460-7. doi: 10.3945/ajcn.115.116939. Epub 2015 Oct 21. PMID 26490495